CLINICAL TRIAL: NCT01864018
Title: Phase 1/2 Trial of Ixazomib in Combination With Cyclophosphamide and Dexamethasone in Patients With Previously Untreated Symptomatic Multiple Myeloma or Light Chain Amyloidosis
Brief Title: Ixazomib With Cyclophosphamide and Dexamethasone in Patients With Previously Untreated Symptomatic Multiple Myeloma or Light Chain Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1382; NCI-2013-01042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16009 (Other: Sponsor Protocol Number); MC1382 (Other: Mayo Clinic); 13-000414 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Amyloidosis; Plasma Cell Myeloma
MeSH Terms: conditions — Amyloidosis; Multiple Myeloma | interventions — Cyclophosphamide; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixazomib citrate, cyclophosphamide, dexamethasone) (Experimental): INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial studies the side effects and the best dose of cyclophosphamide when given together with ixazomib citrate and dexamethasone in treating patients with previously untreated symptomatic multiple myeloma or light chain amyloidosis. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cyclophosphamide together with ixazomib citrate and dexamethasone may be a better treatment for multiple myeloma or light chain amyloidosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of cyclophosphamide that can be combined with ixazomib citrate (ixazomib) and dexamethasone in patients with previously untreated symptomatic multiple myeloma (MM). (Phase I Cohort A) II. To determine the complete plus very good partial response rate (>= VGPR) of ixazomib, used in combination with cyclophosphamide and dexamethasone in patients with previously untreated symptomatic MM. (Phase II Cohort A) III. To determine the hematologic response rate of ixazomib, used in combination with cyclophosphamide and dexamethasone in patients with previously untreated light chain amyloidosis. (Phase II Cohort B)

SECONDARY OBJECTIVES:

I. To determine the progression free survival and overall survival among patients with previously untreated symptomatic MM following treatment with ixazomib in combination with cyclophosphamide and dexamethasone followed by ixazomib maintenance till progression. (Cohort A) II. To determine the toxicities associated with ixazomib in combination with cyclophosphamide and dexamethasone in patients with previously untreated symptomatic MM. (Cohort A) III. To determine the organ response rate of ixazomib, used in combination with cyclophosphamide and dexamethasone in patients with previously untreated light chain amyloidosis. (Cohort B) IV. To determine the progression free survival and overall survival among patients with previously untreated light chain amyloidosis following treatment with ixazomib in combination with cyclophosphamide and dexamethasone followed by Ixazomib maintenance till progression. (Cohort B) V. To determine the toxicities associated with ixazomib in combination with cyclophosphamide and dexamethasone in patients with previously untreated light chain amyloidosis. (Cohort B)

TERTIARY OBJECTIVES:

I. To examine the pharmacokinetics of ixazomib when used in combination with cyclophosphamide and dexamethasone. (Cohort A) II. To assess the incidence of neurotoxicity using patient completed questionnaires. (Cohort A)

OUTLINE: This is a phase I, dose-escalation study of cyclophosphamide followed by a phase II study.

INDUCTION THERAPY: Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I ONLY:
* COHORT A: multiple myeloma
* COHORT B: biopsy proven light chain amyloidosis with organ involvement requiring therapy
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 75000/mm^3
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* COHORT B ONLY: alkaline phosphatase =< 750 U/L
* COHORT B ONLY: N-terminal pro b-type natriuretic peptide (NT-ProBNP) < 7500 ng/dL
* Prior therapy for the treatment of solitary plasmacytoma is permitted, but > 14 days should have elapsed from the last day of radiation; NOTE: prior therapy with clarithromycin, dehydroepiandrosterone (DHEA), anakinra, pamidronate or zoledronic acid is permitted; any additional agents not listed must be approved by the principal investigator
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* COHORT B ONLY: serum immunoglobulin free light chain >= 5 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Previously untreated
* Provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures as suggested by the study

  * Female patients: if they are of childbearing potential, agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to return to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma only
* Prior cytotoxic chemotherapy or corticosteroids for the treatment of multiple myeloma; NOTE: prior corticosteroid use for the treatment of non-malignant disorders is permitted
* Diagnosed or treated for another malignancy =< 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; NOTE: patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 3 on clinical examination or grade 2 with pain during the screening period
* Major surgery =< 14 days prior to study registration
* Systemic treatment with strong CYP3A4 inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, Gingko biloba, St. John?s wort) =< 14 days prior to registration
* Evidence of current uncontrolled cardiovascular conditions (New York Heart Association [NYHA] class III or IV), including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction within the past 6 months; Note: prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Radiotherapy =< 14 days prior to registration; NOTE: if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Any serious medical or psychiatric illness that could, in the investigator?s opinion, potentially interfere with the completion of treatment according to this protocol
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grading, in the absence of antidiarrheals
* Participation in clinical trials with other investigational agents not included in this trial, =< 30 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Muchtar E, Gertz MA, LaPlant BR, Buadi FK, Leung N, O'Brien P, Bergsagel PL, Fonder A, Hwa YL, Hobbs M, Helgeson DK, Bradt EE, Gonsalves W, Lacy MQ, Kapoor P, Siddiqui M, Larsen JT, Warsame R, Hayman SR, Go RS, Dingli D, Kourelis TV, Dispenzieri A, Rajkumar SV, Kumar SK. Phase 2 trial of ixazomib, cyclophosphamide, and dexamethasone for previously untreated light chain amyloidosis. Blood Adv. 2022 Sep 27;6(18):5429-5435. doi: 10.1182/bloodadvances.2022007781. PMID 35737873
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase I participants are grouped with the phase II, cohort A participants because they were grouped in the published manuscript
Groups:
- Phase I/II, Cohort A: Patients with Multiple Myeloma>
  > INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies
- Phase II, Cohort B: Patients with biopsy proven light chain amyloidosis with organ involvement> requiring therapy>
  > INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B
Started | 51 | 36
Accrued During Phase I | 10 | 0
Accrued During Phase II | 41 | 36
Completed | 48 | 35
Not Completed | 3 | 1
Not completed — Ineligible | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B | Total
Number analyzed (Participants) | 48 | 35 | 83
Age, Continuous [Median (Full Range); unit: years] | 64.5 [41 to 88] | 67 [38 to 78] | 65 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 46 | 35 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 35 | 83
ECOG Performance Status [Count of Participants; unit: Participants] — Grade 0 - Fully active, able to carry on all pre-disease performance without restriction> Grade 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work> Grade 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 25 | 16 | 41
    1 | 19 | 17 | 36
    2 | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated (MTD) Dose of Cyclophosphamide With Ixazomib and Dexamethasone (Phase I)
Description: Will be defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least 1/3 of patients, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: At 28 days
Population: The 10 patients accrued to the phase I portion of the study were analyzed to determine the maximum tolerated dose of ixazomib with cyclophosphamide and dexamethasone
Measure: Number; unit: mg weekly
Groups:
- Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone): INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.> >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies
Arm/Group | Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone)
Number analyzed (Participants) | 10
mg weekly
  MTD of ixazomib | 4
  MTD of dexamethasone | 40

2. Primary Outcome: Percentage of Patients With Complete Response or Very Good Partial Response (Phase II, Cohort A)
Description: The percentage of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: Up to 48 weeks
Population: Includes only eligible patients in phase II, cohort A
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone)
Number analyzed (Participants) | 48
percentage of participants | 35 [22 to 50]

3. Primary Outcome: Rate of Complete Response, Very Good Partial Response, or Partial Response (Phase II, Cohort B)
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated.
Time Frame: Up to 48 weeks
Population: Includes only patients with biopsy proven light chain amyloidosis with organ involvement>> requiring therapy at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone): INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>> >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>>
  >> Cyclophosphamide: Given PO>>
  >> Dexamethasone: Given PO>>
  >> Ixazomib Citrate: Given PO>>
  >> Laboratory Biomarker Analysis: Correlative studies>>
  >> Pharmacological Study: Correlative studies>>
  >> Quality-of-Life Assessment: Ancillary studies>>
  >> Questionnaire Administration: Ancillary studies
Arm/Group | Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone)
Number analyzed (Participants) | 35
percentage of participants | 63 [45 to 79]

4. Secondary Outcome: Number of Patients Experiencing a Grade 3 or Greater Adverse Event at Least Possibly Related to Treatment as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. A grade 3 event is one that is severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B
Number analyzed (Participants) | 48 | 35
Participants | 36 | 16

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The distribution of PFS will be estimated using the method of Kaplan Meier.
Time Frame: Time from registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I/II, Cohort A: Patients with multiple myeloma> > INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies>
  >>
  >
  >> Patient has multiple myeloma at baseline
- Phase II, Cohort B: Patients with biopsy proven light chain amyloidosis with organ involvement requiring therapy>
  >
  > INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies>
  >>
  >
  >> Patient has light chain amyloidosis at baseline
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B
Number analyzed (Participants) | 48 | 35
months | NA [31.3 to NA] — Median and upper 95% CI PFS was not reached due to the low number of progressions (11) | NA [39.6 to NA] — Median and upper 95% CI PFS was not reached due to the low number of progressions (5)

6. Secondary Outcome: Survival Time
Description: The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II, Cohort B: Patients with biopsy proven light chain amyloidosis with organ involvement requiring therapy> > INDUCTION THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15 and cyclophosphamide PO and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> MAINTENANCE THERAPY: Patients receive ixazomib citrate PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  >>
  >
  >> Cyclophosphamide: Given PO>
  >>
  >
  >> Dexamethasone: Given PO>
  >>
  >
  >> Ixazomib Citrate: Given PO>
  >>
  >
  >> Laboratory Biomarker Analysis: Correlative studies>
  >>
  >
  >> Pharmacological Study: Correlative studies>
  >>
  >
  >> Quality-of-Life Assessment: Ancillary studies>
  >>
  >
  >> Questionnaire Administration: Ancillary studies>
  >>
  >
  >> Patient has light chain amyloidosis at baseline
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B
Number analyzed (Participants) | 48 | 35
months | NA [NA to NA] — Median and 95% CI PFS was not reached due to the low number of deaths (2) | NA [NA to NA] — Median and 95% CI PFS was not reached due to the low number of deaths (7)

7. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters
Description: Will be estimated using noncompartmental analysis methods. The plasma PK parameters calculated for individual plasma ixazomib concentration-time data will include, but are not limited to: peak concentration, time to first maximum plasma concentration, and area under the curve. PK parameters will be summarized using descriptive statistics.
Time Frame: Post-dose, 1 and 4 hours on day 1, pre-dose on days 8, 15, and 22, and day 1 of course 2
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quality of Life, as Assessed by the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity Questionnaire
Description: Patients will be evaluated by overall score at each time point and changes over time will be calculated. These measures will be correlated with outcome using Fisher's exact test and Kaplan-Meier methods where appropriate.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Primary Outcome: Maximum Tolerated (MTD) Dose of Cyclophosphamide (Phase I)
Description: as for outcome 1
Time Frame: At 28 days
Population: as for outcome 1
Measure: Number; unit: mg/m² weekly
Arm/Group | Treatment (Ixazomib Citrate, Cyclophosphamide, Dexamethasone)
Number analyzed (Participants) | 10
mg/m² weekly | 400

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Phase I/II, Cohort A; Phase II, Cohort B: Questionnaire Administration: Ancillary studies
Arm/Group | Phase I/II, Cohort A | Phase II, Cohort B
All-Cause Mortality (participants affected / at risk) | 2/48 | 7/35
Serious Adverse Events (participants affected / at risk) | 16/48 | 15/35
Other Adverse Events (participants affected / at risk) | 48/48 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II, Cohort A (N=48) | Phase II, Cohort B (N=35)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 2 (2)
Weight gain (Investigations) | 1 (12) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II, Cohort A (N=48) | Phase II, Cohort B (N=35)
Anemia (Blood and lymphatic system disorders) | 14 (29) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 1 (5) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (4) | 0 (0)
Cataract (Eye disorders) | 1 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 36 (179) | 25 (68)
Diarrhea (Gastrointestinal disorders) | 29 (115) | 15 (48)
Duodenal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 29 (138) | 22 (66)
Vomiting (Gastrointestinal disorders) | 12 (17) | 6 (11)
Edema limbs (General disorders) | 1 (2) | 6 (10)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 47 (546) | 32 (221)
Pain (General disorders) | 1 (4) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (4) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (3) | 1 (5)
CD4 lymphocytes decreased (Investigations) | 5 (5) | 0 (0)
Creatinine increased (Investigations) | 10 (25) | 15 (138)
Lymphocyte count decreased (Investigations) | 42 (296) | 9 (40)
Lymphocyte count increased (Investigations) | 5 (8) | 2 (2)
Neutrophil count decreased (Investigations) | 29 (138) | 2 (3)
Platelet count decreased (Investigations) | 31 (86) | 11 (25)
White blood cell decreased (Investigations) | 42 (230) | 6 (8)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (9) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 9 (24) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 35 (361) | 19 (91)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (10) | 8 (18)
Libido decreased (Psychiatric disorders) | 1 (9) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19 (34) | 11 (70)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (12) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT01864018/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT01864018/ICF_001.pdf